CLINICAL TRIAL: NCT05006339
Title: The Use of Remote Monitoring for Orthodontic Retention Review: A Randomised Controlled Trial
Brief Title: The Use of Remote Monitoring for Orthodontic Retention Review
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X20-0358
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Orthodontic Relapse
Keywords: Orthodontic retention; Orthodontic relapse; Dental monitoring; Remote monitoring; AI supported remote orthodontic monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Monitoring (Experimental): Orthodontic retention review via dental monitoring only
  Interventions: Device: Dental Monitoring
- Clinic Review (Active Comparator): Orthodontic retention review via in-office visits as per routine care
  Interventions: Other: Clinic Review

INTERVENTIONS:
Device: Dental Monitoring — Patients in this arm are not required to attend in-office retention appointments except if they have any problems with their retainers and when data collection is necessary. Instead they are required to submit scans of their teeth through the DM mobile application at the designated intervals.
  Arms: Dental Monitoring
Other: Clinic Review — Patients in this arm are required to attend in clinic appointments for their retention review
  Arms: Clinic Review

SUMMARY:
To assess whether using retainers and an artificial intelligence supported remote monitoring system maintains a more stable orthodontic treatment result than using retainers with in-office review appointments.

DETAILED DESCRIPTION:
The amount and nature of relapse are unpredictable and natural changes in the dentition are life-long. Although some patients were shown to remain stable despite not wearing retainers, research is unable to provide predictors for identifying those patients and therefore we have to treat all patients as if they have the potential to relapse long term.

Following the results of long-term retrospective studies, there has been a gradual change of practice from prescribing retainers for 1-2 years to long-term retention. This is a significant burden on patients, clinicians and the health system as long term review and maintenance of retainers are required from both parties.

Although some studies showed compliance with the use of orthodontic retainers correlated with factors such as gender, age and type of retainer, one of the main reasons for non-compliance with removable retainers was shown to be just forgetting to wear them. Patient compliance is also needed in attending follow-up appointments for review of fit and intactness of retainers as well as calculus build-up that may be present around fixed lingual wires.

Long term review is also needed to protect patients from any side effects from broken or distorted fixed retainers. This is not common, yet when it happens its side effects can be deleterious. Since patients do not always realise these side effects on time, damage may range from simple malalignment of teeth to having roots of teeth come out of bone creating periodontal and aesthetic consequences.

Attending review appointments could be inconvenient for both patients and parents as they need to take time off of school and work.

There are currently no studies on the efficacy of DM as a tool to monitor orthodontic retention patients. Therefore, this project can shed light on whether the use of DM is an acceptable or more effective way of monitoring patients wearing retainers than traditional in-office orthodontic visits. The results of this study could also help guide clinicians regarding the most effective retention regime using remote monitoring systems. The study will also compare the costs of in-office retainer checks and remote monitoring of retainers, If the results of this study show DM is better, or comparable to, clinical review appointments and it less costly and more convenient, DM may be utilised for patients in the public system freeing chair-time for patients waiting for treatment on the public orthodontic waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the trial and comply with the retention regime and able to follow instructions
* Permanent dentition
* Good general health
* Good oral hygiene and good periodontal health
* Owning or having access to a mobile/smart phone compatible with Dental monitoring application (DM app is available for use on all iOS and Android devices)

Exclusion Criteria:

* Patients with

  * Congenital anomalies or craniofacial syndromes
  * Poor oral hygiene and poor periodontal health
  * Missing teeth & teeth with poor enamel quality
* Patients that were treated with orthognathic surgery
* Patients that are unwilling or unable to follow the instructions provided

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Orthodontic treatment stability - Little's Irregularity Index | 4 years
  The sum of the linear displacements of five labial segment contact point in a labiolingual direction
Orthodontic treatment stability - Spacing if present | 4 years
  The sum of the linear distances between contact points of teeth that have space between them
Orthodontic treatment stability - Inter-canine width | 4 years
  Distance between the cusp tips of right and left canines
Orthodontic treatment stability - Inter-molar width | 4 years
  Distance between the mesiobuccal cusp tips of the right and left first permanent molars
Orthodontic treatment stability - Overjet | 4 years
  The maximum distance between the upper incisors edge and the lower incisal labial surface
Orthodontic treatment stability - Overbite | 4 years
  The maximum vertical overlap between the upper and lower incisors with the models in maximal intercuspation

SECONDARY OUTCOMES:
Retainer failure | 4 years
  Retainer failure identification, yes or no
Retainer failure identification time | 4 years
  Retainer failure identification duration, in number of days
Retainer problems - compliance | 4 years
  Retainer compliance measured with fit of retainer - space in mm between retainer and teeth
Oral Health Assessment - Cavity presence if any | 4 years
  Identification of cavities
Oral health assessment - Gingivitis if any | 4 years
  Identification of gingivitis
Patient satisfaction | 4 years
  Satisfaction with the 2 protocols of retention review using Likert scale questionnaires that have 5 answer options ranging from "strongly agree" to "strongly disagree". Different questions have positive/negative outcomes with either end of the scale.
Cost effectiveness | 4 years
  Total cost of both systems

CONTACTS AND LOCATIONS:
Overall Officials: Oyku Dalci, DDS, PhD, Principal Investigator — Sydney Local Health District, The University of Sydney
Locations (1):
- Sydney Dental Hospital, Surry Hills, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No